CLINICAL TRIAL: NCT00341952
Title: Interdisciplinary Case-Control Study of Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998022; OH98-C-N022
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Case-Control Study; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: individuals diagnosed with incident, first primary non-Hodgkin lymphoma
- Controls: individuals identified in the same geographical areas without non-Hodgkin lymphoma or othercancers

SUMMARY:
Non-Hodgkin's lymphoma (NHL) incidence rates have risen three percent per year in the U.S. for four decades. Mortality from NHL has risen 1.6 percent, compared with 0.2 percent for all cancers combined. This epidemic curve appears in both sexes and around the world, suggesting the possibility of an etiologic agent increasing in prevalence in the general environment. Recent research has identified several possible candidates including pesticides, other organochlorines, drinking water nitrates, and sunlight. There is an urgent need to evaluate whether these common exposures are contributing to the rapid rise in NHL, and to investigate other hypothesized risk factors such as viruses, medical conditions, hair dye use, and genetic factors. The purpose of this study is to examine the contribution to NHL risk of these important environmental, occupational, viral, medical, and personal exposures, and to pursue important leads emerging from on-going NHL research. This multidisciplinary, population-based case-control study will involve personal interviews to collect information on demographics, residential history, pesticide use, and occupational exposures; self-administered questionnaires to collect information on diet, family and medical history, and other exposures; tap water and carpet dust sampling to collect information on nitrate and pesticide exposures; and blood sampling for measurements of compounds in the serum, antibodies to viruses, and examination of genetic polymorphisms.

DETAILED DESCRIPTION:
Non-Hodgkin's lymphoma (NHL) incidence rates have risen three percent per year in the U.S. for four decades. Mortality from NHL has risen 1.6 percent, compared with 0.2 percent for all cancers combined. This epidemic curve appears in both sexes and around the world, suggesting the possibility of an etiologic agent increasing in prevalence in the general environment. Recent research has identified several possible candidates including pesticides, other organochlorines, drinking water nitrates, and sunlight. There is an urgent need to evaluate whether these common exposures are contributing to the rapid rise in NHL, and to investigate other hypothesized risk factors such as viruses, medical conditions, hair dye use, and genetic factors. The purpose of this study is to examine the contribution to NHL risk of these important environmental, occupational, viral, medical, and personal exposures, and to pursue important leads emerging from on-going NHL research. This multidisciplinary, population-based case-control study will involve personal interviews to collect information on demographics, residential history, pesticide use, and occupational exposures; self-administered questionnaires to collect information on diet, family and medical history, and other exposures; tap water and carpet dust sampling to collect information on nitrate and pesticide exposures; and blood sampling for measurements of compounds in the serum, antibodies to viruses, and examination of genetic polymorphisms.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Women and men residing in the areas served by the four SEER registries.

Individuals between the ages of 20 and 74 (ages between 20 and 64 must live in households with telephones).

Individuals who have a first primary diagnosis of NHL after April 1, 1998 to July 1, 1998.

Individuals must be HIV negative.

EXCLUSION CRITERIA:

Individuals must not be previously diagnosed with NHL.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of participating SEER registries
Sampling Method: Probability Sample
Enrollment: 2378 (Actual)
Dates: Start 1998-04-15; Primary Completion 2007-04-17 (Actual); Study Completion 2007-04-17 (Actual)

PRIMARY OUTCOMES:
No intervention. Observational study compares cases and controls. | at the time of enrollment
  non-Hodgkin lymphoma cases versus controls

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Rothman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - University of Iowa, Iowa City, Iowa
  - Wayne State University Hutzel Hospital, Detroit, Michigan
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Gridley G, McLaughlin JK, Ekbom A, Klareskog L, Adami HO, Hacker DG, Hoover R, Fraumeni JF Jr. Incidence of cancer among patients with rheumatoid arthritis. J Natl Cancer Inst. 1993 Feb 17;85(4):307-11. doi: 10.1093/jnci/85.4.307. PMID 8426374
- [Background] Cantor KP, Blair A, Everett G, VanLier S, Burmeister L, Dick FR, Gibson RW, Schuman L. Hair dye use and risk of leukemia and lymphoma. Am J Public Health. 1988 May;78(5):570-1. doi: 10.2105/ajph.78.5.570. PMID 3354743
- [Background] Bentham G. Association between incidence of non-Hodgkin's lymphoma and solar ultraviolet radiation in England and Wales. BMJ. 1996 May 4;312(7039):1128-31. doi: 10.1136/bmj.312.7039.1128. PMID 8620128